CLINICAL TRIAL: NCT00404560
Title: Screening Protocol for Detection and Characterization of Infections and Infection Susceptibility
Brief Title: Detection and Characterization of Infections and Infection Susceptibility
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070033; 07-I-0033
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-06

CONDITIONS: Immune Deficiencies
Keywords: Primary Immune Deficiency; Autoimmune; Genetic Defects; Immune Defects; Infection Susceptibility; Recurrent Infections; Immune Disorders; Immune Defects of Phagocytes; Unusual, Chronic Bacterial, Mycobacterial, and Fungal Infections
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Reinfection; Immune System Diseases; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy blood relatives: relatives not ill with a known or suspected infection susceptibility syndrome
- Patients: patients who either have, or are suspected of having, an infection or infection susceptibility in order to further characterize such conditions

SUMMARY:
This screening study will examine the causes of immune disorders affecting white blood cells, which defend against infections and will try to develop better means of diagnosis and treatment of these immune disorders. This is a 2 visit screening study and patients determined to be of interest for additional study or treatment will be asked to provide consent for enrollment into an appropriate NIH follow up study. This study does not cover the cost of the first visit to NIH for travel or lodgings but does cover the subsequent visit if there is one. A financial assessment may determine if the patient is eligible for financial assistance. This study does not enroll children under the age of 2.

Patients known to have or suspected of having increased susceptibility to infections and their blood relatives may be eligible for this study, at the discretion of the principal investigator. Patients and family members may undergo the following procedures:

* Personal and family medical history.
* Physical examination and blood and urine tests.
* Studies of breathing function (pulmonary function testing)
* Dental examination.
* Eye examination.
* Genetic Testing
* Stored specimens for future analysis
* Microscopic examination of saliva, wound drainage or tissues removed for medical reasons for cell, hormone or DNA studies.

In addition, patients will be asked to obtain permission for investigators to obtain their medical records, previous test results, or radiographic studies prior to the first visit. Patients will be asked to undergo imaging studies, such as a chest X-ray, CT scan or MRI scan.

DETAILED DESCRIPTION:
This screening study is designed to evaluate patients with suspected or identified recurrent or unusual infections and their family members for clinical and in vitro correlates of exposure and susceptibility. It will allow for up to 2 visits to obtain blood, urine, saliva, stool, skin biopsy, or wound drainage from such patients or their family members for research studies related to understanding the nature of the infection as well as the genetic and biochemical bases of these diseases. Patients determined by initial evaluation to be of interest for additional study or treatment will be asked to provide consent for enrollment into an appropriate NIH follow-up study. The present study will enroll up to 2000 patients and family members over the next 25 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS:

* Patients known to have, or suspected of having an infection susceptibility and their healthy blood relatives will be eligible for enrollment.
* Participants must be over 1 month of age. There will be no limit as to sex, race or disability.
* Patients must have a primary physician outside of the NIH and may be required to submit a letter from their physician that documents their relevant health history.
* The participant or the participant's guardian will be willing and capable of providing informed consent after initial counseling by clinical staff. Separate consent forms for all interventional procedures will be obtained after explanation of the specific procedure.
* Patients and relatives must agree to have blood and tissue stored for future studies of the immune system and/or other medical conditions.
* Patients and relatives may be concurrently enrolled on other protocols as long as the Principal Investigator is informed.
* The patient must be enrolled on this protocol to have relatives enrolled.

The patient and patient relative cohorts will include the following special populations:

* Children: Children are included in this study because immune defects may present in early childhood, and early diagnosis or characterization may benefit subjects. Children who do not meet the age and weight criteria for care at the Clinical Center, may have sample collection only.
* Decisionally impaired adults: Patients and patient relatives will be able to provide informed consent for themselves or, if they lack the capacity to provide informed consent, the study team will obtain consent from the legally authorized representative. Patients with underlying immune disorders, autoimmune phenomena or severe infections may sometimes present with delirium, encephalopathy, or coma and are therefore unable to provide informed consent. Excluding patients who are unable to provide consent could adversely impact patient access to medical therapy at the NIH as well as adversely impact research recruitment. Excluding patients unable to provide consent would also essentially prohibit us from evaluating patients at higher risk for adverse outcomes and therefore skew our understanding of disease. Similarly, enrolled patient subjects who lose the ability to provide ongoing consent during study participation may continue in the study. The risks and benefits of participation for subjects unable to consent should be identical to those described for less vulnerable patients.

EXCLUSION CRITERIA:

1. A well understood acquired abnormality which leads to infection susceptibility, such as HIV, cytotoxic chemotherapy, or active malignancy may be adequate explanation for the infection diathesis. These may be grounds for exclusion if, in the opinion of the investigators, the presence of such disease process interferes significantly with evaluation (applicable to patients and their blood relatives).
2. Severe or uncommon infections or syndromes often require highly specialized teams and institutions. Some referred cases will not be able to be handled appropriately at the NIH and may be deemed ineligible for admission, as determined by the Principal Investigator.
3. Pregnancy

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-01-02 (Actual)

PRIMARY OUTCOMES:
determination of a discrete diagnosis of an infecting agent, an underlying susceptibility trait, or both. | upon diagnosis or after the second visit
  patients determined to have a diagnosis or syndrome that requires further study at the NIH will be asked to provide consent for enrollment into an appropriate study for further diagnosis and/or treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this study for future research as follows:@@@-Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC).@@@-De-identified or identified data with approved outside collaborators under appropriate agreements.@@@-Data sharing may be complicated or limited in certain cases by contractual obligations or agreements with outside collaborators, such as cooperative research and development agreements, clinical trial agreements, other restraints, etc.
Supporting Information: SAP
Time Frame: IPD and supporting information will be available after completion of the study. No end date.
Access Criteria: Data will be shared through:@@@-BTRIS (automatic for activities in the NIH CC).@@@-Approved outside collaborators under appropriate individual agreements.@@@-Publication and/or public presentations.@@@-Data might be shared before publication.@@@-The PI will review all requests for sharing data.

REFERENCES:
- [Background] Chien WW, Leiding JW, Hsu AP, Zalewski C, King K, Holland SM, Brewer C. Auditory and vestibular phenotypes associated with GATA3 mutation. Otol Neurotol. 2014 Apr;35(4):577-81. doi: 10.1097/MAO.0000000000000238. PMID 24622013
- [Background] Saijo T, Chen J, Chen SC, Rosen LB, Yi J, Sorrell TC, Bennett JE, Holland SM, Browne SK, Kwon-Chung KJ. Anti-granulocyte-macrophage colony-stimulating factor autoantibodies are a risk factor for central nervous system infection by Cryptococcus gattii in otherwise immunocompetent patients. mBio. 2014 Mar 18;5(2):e00912-14. doi: 10.1128/mBio.00912-14. PMID 24643864
- [Background] Spinner MA, Sanchez LA, Hsu AP, Shaw PA, Zerbe CS, Calvo KR, Arthur DC, Gu W, Gould CM, Brewer CC, Cowen EW, Freeman AF, Olivier KN, Uzel G, Zelazny AM, Daub JR, Spalding CD, Claypool RJ, Giri NK, Alter BP, Mace EM, Orange JS, Cuellar-Rodriguez J, Hickstein DD, Holland SM. GATA2 deficiency: a protean disorder of hematopoiesis, lymphatics, and immunity. Blood. 2014 Feb 6;123(6):809-21. doi: 10.1182/blood-2013-07-515528. Epub 2013 Nov 13. PMID 24227816
- [Derived] West RR, Hsu AP, Holland SM, Cuellar-Rodriguez J, Hickstein DD. Acquired ASXL1 mutations are common in patients with inherited GATA2 mutations and correlate with myeloid transformation. Haematologica. 2014 Feb;99(2):276-81. doi: 10.3324/haematol.2013.090217. Epub 2013 Sep 27. PMID 24077845
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-I-0033.html